CLINICAL TRIAL: NCT03840876
Title: Supraglottic Jet Oxygenation and Ventilation Via Nasal Approach During Laser Microlaryngeal Surgery for Vocal Polyps Resection
Brief Title: SJOV With WNJ in Microlaryngeal Surgery
Acronym: WNJ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Hui Qiao, Attending Anesthesiologist, Eye & ENT Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WNJ
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Other Complications of Surgical and Medical Procedures
Keywords: Jet Ventilation; Supraglottic; Intranasal; Microlaryngeal Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group J (Experimental): Jet ventilation was achieved via supraglottic jet oxygenation and ventilation with WEI NASAL JET (WNJ).
  Interventions: Device: WEI NASAL JET (WNJ)
- Group I (No Intervention): Patients were ventilated with a small size endotracheal tube.

INTERVENTIONS:
Device: WEI NASAL JET (WNJ) — Jet ventilation was achieved with WEI NASAL JET (WNJ) connected to a manual jet ventilator (Driving pressure: 40 psi, fraction of inspired oxygen: 100% O2, Respiratory rate: 25/min, I/E ratio: 40%)
  Arms: Group J

SUMMARY:
The key to a successful microlaryngoscopy is adequate operative field exposure and illumination. A variety of airway control procedures has been developed to improve operative exposure. A small size endotracheal tube is commonly used. However, some surgeon may suggest a 'no-tube' technique to optimize the surgical field. This study aims to investigate effectiveness and safety of a novel technique by supraglottic jet oxygenation and ventilation (SJOV) via nasal approach to facilitate optimal visualization in laser microlaryngeal surgery for small vocal polyps resection.

DETAILED DESCRIPTION:
The allocation sequence is generated by computer random number generation, and the allocation is placed in sequentially numbered opaque sealed envelopes by a non-investigator. Enrolment and data collection are performed by trained research staff who are not involved in the care of the patients. The treating clinicians are not possible to be blinded to the assignment group, but all other staff involved in both the collection and collation of data, and administration of neurocognitive testing, are blinded to group allocation.

The primary measurement is numerical rating scale (NRS) rated by surgeon according to surgical exposure and visualization. The secondary measurements are operation duration, and Intraoperative pulse oximetry (SpO2), PetCO2.

The continuous variables were expressed as means ± standard deviation (SD) whereas categorical variables were expressed as frequency and percentage for data description.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for laser laryngeal surgery under general anesthesia

Exclusion Criteria:

* Patients with cardiac, pulmonary, hepatic, or renal dysfunction. Patients with nasal disease. Patients with anticipated difficult airway.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Numerical rating scale (NRS) rated by surgeon | Immediately after surgery, the surgeons rated surgical exposure and visualization with NRS only once.
  The surgeons rated surgical exposure and visualization on a numerical rating scale (NRS), ranging from 0 to 10, with 0 defined as the best condition and 10 as the worst.

SECONDARY OUTCOMES:
Operation duration | Immediately after surgery, the duration of the operation was recorded by the investigator.
  Duration of the operation

CONTACTS AND LOCATIONS:
Overall Officials: Wenxian Li, M.D. Ph.D., Study Director — Eye and ENT Hospital of Fudan University
Locations (1):
- Eye, Ear, Nose and Throat Hospital, Shanghai, Shanghai Municipality, China